CLINICAL TRIAL: NCT04478604
Title: The Evaluation of Anxiety and Anxieties Related to Childbirth and Postpartum Period With Childbirth Pain in Last Trimester Pregnant Women
Brief Title: Anxieties Related to Childbirth and Postpartum Period
Acronym: Anxietybirth
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Meltem Ugurlu, Assistant professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: SBUuniversitesi
Record Dates: First submitted 2020-07-16; First posted 2020-07-20 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Childbirth Fear, Anxiety,Birth Pain
Keywords: Pregnancy, Childbirth, Postpartum period, Nursing care
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women: last trimester pregnant women and gave birth in the same hospital
  Interventions: Other: applied forms to pregnant women

INTERVENTIONS:
Other: applied forms to pregnant women
  Other Names: Sociodemographic and Obstetric Features Questionnaire,Fear of Childbirth and Postpartum Anxiety Scale,Spielberger State and Trait Anxiety Inventory

SUMMARY:
The present study aimed to evaluate the relation of labor pain with anxiety and worries about labor and postpartum period in pregnant women in their last trimester.

DETAILED DESCRIPTION:
During pregnancy and after childbirth, women experience many physical, emotional and psychological changes and try to cope with them1. Many women have fear of childbirth and anxiety for various reasons such as uncertainties about labor, labor pain, loss of control and giving birth alone 2,3. Several studies have shown that 12%-31% of the pregnant women experience fear of childbirth 4-6. The sources of worries are usually the possible risk of harm to women themselves or their babies and attitudes and insufficient knowledge of health staff2,6-8. These prenatal worries may lead to pain and restlessness during labor, emergency cesarean section and postpartum affective disorders 1.

Stress experienced during pregnancy affects not only maternal health but also childbirth outcomes (e.g. preterm labor and low birth weight) 9. Anxiety most frequently experienced in the first and last trimesters are not directly associated with obstetric complications; however, it may cause obstetric complications due to the changes it created in the endocrine system1,7,9. Although labor pain can be due to physiological changes such as cervix dilatation and uterus contractions, it may result from psychological factors like stress, anxiety and fear 10. In several studies, the relation between state and trait anxiety scores just before or during childbirth and pain experienced during labor has been evaluated 11,12.

According to the World Health Organization (WHO), the purpose of the antenatal care is to help women to have a positive childbirth experience 13. Positive expectations about childbirth during pregnancy may lead to a positive childbirth experience, while anxiety, fear or negative expectations can create a negative childbirth experience 14. Several studies have shown that antenatal education decreases anxiety and labor pain 15,16.

It is of importance to reveal worries and anxiety experienced by pregnant women during and after childbirth and to evaluate their relationship with labor pain in terms of provision of higher-quality antenatal care and development of more effective coping strategies to deal with these problems. Thereby, women may be more healthy during their pregnancy and have a positive childbirth experience.

This study aimed to determine the relation of labor pain with worries about childbirth and the postpartum period and state-trait anxiety levels in pregnant women in the last trimester.

MATERIAL AND METHODS The study has a descriptive, prospective design and was conducted in the obstetric clinic of a research and education hospital between January and November in 2014. The study population included the pregnant women in their third trimester presenting to the obstetrics outpatient clinic of the hospital at the time of the study and the sample comprised 115 pregnant women planning to give birth in the same hospital. Since five women did not volunteer to participate in the study and since six women gave birth in another hospital, the study was performed with 104 women (90%).

Data collection tools Data were gathered with a sociodemographic and obstetric features questionnaire created by the researchers in light of the literature, 1,11,17 Fear of Childbirth and Postpartum Anxiety Scale (FCPAS), Spielberger State and Trait Anxiety Inventory (STAI) and Visual Analogue Scale (VAS).

Sociodemographic and Obstetric Features Questionnaire The questionnaire was composed of two sections. The first section involved questions about sociodemographic features including age, employment status and education. The second section involved 11 questions about the total number of pregnancies, outcome of the prior pregnancy, experiencing problems during the prior pregnancy, experiencing problems in the current pregnancy and planned mode of childbirth.

Fear of Childbirth and Postpartum Anxiety Scale FCPAS was developed by Kitapçıoğlu et al. in 2007 to determine worries experienced during and after childbirth 1. The scale is composed of ten subscales and 61 items. It is a five-point Likert scale and one corresponds to completely disagree and five totally agree. Some items are scored in the reverse order. The scores for the scale range from zero to ten. The scores 0.00-2.00 are very low, the scores 2.01-4.00 are low, the scores 4.01-6.00 are moderate, the scores 6.01-8.00 are high and the scores 8.01-10.00 are very high18. Cronbach's alpha was reported to 0.95 for the original scale1 and it was found to be 0.96 in the present study.

Spielberger State and Trait Anxiety Inventory STAI was developed by Spielberg et al. in 1970 to measure state and trait anxiety levels of individuals. It was adapted to the Turkish culture by Öner and LeCompte in 198519,20. The inventory is composed of two scales; i.e. state anxiety scale (STAI-State) and trait anxiety scale (STAI-Trait), and each involves 20 items. The former is directed towards determining how individuals feel at a certain moment and under a certain condition, whereas the latter shows how individuals feel in general. STAI is a four-point Likert scale. The total score for the inventory changes between 20 and 80. The scores 0-19 show lack of anxiety, the scores 20-39 mild anxiety, the scores 40-59 moderate anxiety, the scores 60-79 severe anxiety and the score 80 and over 80 very severe anxiety 20.

Visual Analogue Scale VAS was developed by Price et al. in 1983 to measure the severity of pain 21. It is frequently used to determine the severity of pain experienced by women during labor 3,11. Individuals are asked to assign a score for their pain on a 10cm-scale ranging from zero to ten. Zero corresponds to lack of pain and ten corresponds to very severe pain.

Data Collection The women were given information about the aim and methods of the study and their participation in the study had a voluntary basis. Those accepting to participate in the study and planning to give birth in the hospital where this study was conducted were given the data collection tools and requested to complete them by the researcher . It took 15 minutes for each participant to fill them in. The researcher answered the questions asked by the participants during the data collection process. The participants were given the researcher's phone number and asked to call when they came to hospital to give birth. In addition, every day during the study period, the researchers checked whether there were any participants among the women presenting to the hospital to give birth. The pain severity was evaluated by using VAS in the women giving normal birth in the delivery room during the active phase of labor and in the women having cesarean section in the postpartum four hours.

Ethical considerations Ethical approval was obtained from the ethical committee (date of approval: 16.12.2013) and written permission was obtained from the hospital where the study was performed. Written consent was taken from the participants after they were informed about the aim and conduction of the study. The study was carried out in accordance with the Declaration of Helsinki .

Data Analysis Obtained data were analyzed with the SPSS for Windows 16.0 (IBM Corporation Armonk, New York, USA). Kolmogorov Smirnov test was used to determine whether the data about continuous variables were normally distributed. Numbers, percentages, median and mean ±standard deviation were used for descriptive statistics. Cronbach's alpha coefficient was determined. For comparative statistics, t test, one-way analysis of variance, Kruskal Wallis test and Mann Whitney U test were utilized. The relation between two continuous variables was analyzed with Spearman correlation test. The statistical significance was set at 0.05 for all the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Having no major complication related to pregnancy
* Being last trimester
* Ability to read and write in Turkish,
* Volunteering to participate in the study
* Planning give birth in the same hospital

Exclusion Criteria:

* Unable to read or write in Turkish
* Being in the last trimester
* Changing the hospital for giving birth.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Last trimester pregnant women with have no major complications
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2014-11-15 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Fear of Childbirth and Postpartum Anxiety Scale | in the third trimester of pregnancy (between the 28-40 gestational week)
  The questionnaire was composed of two sections. The first section involved questions about sociodemographic features including age, employment status and education. The second section involved 11 questions about the total number of pregnancies, outcome of the prior pregnancy, experiencing problems during the prior pregnancy, experiencing problems in the current pregnancy and planned mode of childbirth.

SECONDARY OUTCOMES:
Spielberger State and Trait Anxiety Inventory | in the third trimester of pregnancy (between the 28-40 gestational week)
  STAI was developed by Spielberg et al. in 1970 to measure state and trait anxiety levels of individuals. It was adapted to the Turkish culture by Öner and LeCompte in 198519,20. The inventory is composed of two scales; i.e. state anxiety scale (STAI-State) and trait anxiety scale (STAI-Trait), and each involves 20 items. The former is directed towards determining how individuals feel at a certain moment and under a certain condition, whereas the latter shows how individuals feel in general. STAI is a four-point Likert scale. The total score for the inventory changes between 20 and 80. The scores 0-19 show lack of anxiety, the scores 20-39 mild anxiety, the scores 40-59 moderate anxiety, the scores 60-79 severe anxiety and the score 80 and over 80 very severe anxiety 20.
Visual Analogue Scale | in the active phase of labor and within the first 4 hours after cesarean delivery
  VAS was developed by Price et al. in 1983 to measure the severity of pain 21. It is frequently used to determine the severity of pain experienced by women during labor 3,11. Individuals are asked to assign a score for their pain on a 10cm-scale ranging from zero to ten. Zero corresponds to lack of pain and ten corresponds to very severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Meltem Uğurlu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Curzik D, Jokic-Begic N. Anxiety sensitivity and anxiety as correlates of expected, experienced and recalled labor pain. J Psychosom Obstet Gynaecol. 2011 Dec;32(4):198-203. doi: 10.3109/0167482X.2011.626093. Epub 2011 Oct 31. PMID 22039971
- [Background] Tugut N, Tirkes D, Demirel G. Preparedness of pregnant women for childbirth and the postpartum period: their knowledge and fear. J Obstet Gynaecol. 2015 May;35(4):336-40. doi: 10.3109/01443615.2014.960375. Epub 2014 Sep 29. PMID 25265338
- [Background] Laursen M, Hedegaard M, Johansen C; Danish National Birth Cohort. Fear of childbirth: predictors and temporal changes among nulliparous women in the Danish National Birth Cohort. BJOG. 2008 Feb;115(3):354-60. doi: 10.1111/j.1471-0528.2007.01583.x. PMID 18190372
- [Background] Hildingsson I, Nilsson C, Karlstrom A, Lundgren I. A longitudinal survey of childbirth-related fear and associated factors. J Obstet Gynecol Neonatal Nurs. 2011 Sep-Oct;40(5):532-43. doi: 10.1111/j.1552-6909.2011.01274.x. PMID 22273410